CLINICAL TRIAL: NCT06081517
Title: Evaluating Disparities in Precision Oncology: An Observational Trial in the Context of a Real-World Academic Practice Model
Brief Title: Evaluating Disparities in Precision Oncology
Acronym: EDPO
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Bryan Schneider, Assistant Professor of Clinical Medicine, Indiana University
Other Study IDs: CTO-IUSCCC-0819
Record Dates: First submitted 2023-08-23; First posted 2023-10-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Cancer; Advanced Cancer
Keywords: Precision Medicine; Disparities
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Social Determinants of Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood will be collected for a research grade genome wide association scan using Illumina's Ex Platform to determine ancestry
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Black patients with advanced cancer
  Interventions: Behavioral: Social Determinants of Health and toxicity questionnaires
- Non Black patients with advanced cancer
  Interventions: Behavioral: Social Determinants of Health and toxicity questionnaires

INTERVENTIONS:
Behavioral: Social Determinants of Health and toxicity questionnaires — Collect detailed clinical, and social data from patients to identify significant contributors of disparate survival and toxicity outcomes.

SUMMARY:
This is a non-randomized observational trial designed to collect detailed clinical, social determinant, and genomic data from patients enrolled in molecular oncology tumor boards across four comprehensive cancer centers.

DETAILED DESCRIPTION:
This study proposes an innovative approach leveraging the molecular tumor boards across four comprehensive cancer centers, where real- world, diverse patients with metastatic cancer are seen receiving a broad scope of therapies in the context of precision medicine. The study plans to collect detailed clinical, social, and genomic data from patients to identify significant contributors of disparate survival and toxicity outcomes for patients with metastatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent and HIPAA authorization
2. Patients must be ≥ 18 years old at the time of consent
3. Patients planning to undergo molecular testing as part of their routine cancer care

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those with cancers being referred for molecular testing through their site's precision genomics program.
Sampling Method: Non-Probability Sample
Enrollment: 10600 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Compare Overall Survival between Black patients and White patients (self-reported race) with advanced cancer | through study completion (i.e. death, lost to follow up, or withdraw)-up to 5 years
Compare rate of new onset or worsening therapy- induced peripheral neuropathy (TIPN) between Black patients and White patients with advanced cancer prospectively exposed to a taxane | through study completion (i.e. death, lost to follow up, or withdraw)-up to 5 years

SECONDARY OUTCOMES:
Compare efficacy based on duration on therapy (DOT) between Black and White patients with advanced cancer (using self-reported race and percentage African ancestry) | From baseline to end of treatment (i.e. up to 2 years)
Assess the significance of key attributes (tumor genomics, clinical demographics, SDoH, access, and the intersection of tumor biology and drug impact) on efficacy, and survival outcomes | Baseline
Assess the significance of key attributes (clinical demographics, SDoH, host genomics and prior therapy exposures) on therapy-induced neuropathy | through study completion (i.e. death, lost to follow up, or withdraw)-up to 5 years
Assess the impact of toxicity as measured by dose reductions or dose cessations attributed to TIPN from chart review measured as RDI, a function of the ratio of received to intended doses, and thus accounts for differences in drugs or time of therapy | through study completion (i.e. death, lost to follow up, or withdraw)-up to 5 years
Evaluate for differences in the impact of neuropathy between Black and White cancer patients on change in patient-reported QoL | through study completion (i.e. death, lost to follow up, or withdraw)-up to 5 years
Compare the rate of checkpoint inhibitor -induced immune -related adverse events (irAEs) between White and Black patients | through study completion (i.e. death, lost to follow up, or withdraw)-up to 5 years
Compare the rate of cardiotoxic therapy -induced heart failure between White and Black patients | through study completion (i.e. death, lost to follow up, or withdraw)-up to 5 years
Compare the rate of drug -induced hypertension between White and Black patients | through study completion (i.e. death, lost to follow up, or withdraw)-up to 5 years
Compare utility of precision genomic information defined by the percentage of patients receiving results, screened for or enrolled on a genomically-directed clinical trial, and receiving a targeted therapy between White and Black patients | through study completion (i.e. death, lost to follow up, or withdraw)-up to 5 years
Compare the differences in prevalence of level 1/2 actionable mutations, prior lines of therapy, receipt of a genomically matched therapy and receipt of an FDA-approved drug between Black and White patients | through study completion (i.e. death, lost to follow up, or withdraw)-up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bryan P Schneider, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana, United States